CLINICAL TRIAL: NCT05286242
Title: Evaluating the Immune Response to COVID19 Vaccination in Immunodeficient Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Robert Leet and Clara Guthrie Patterson Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2000029889; 2U19AI089992-11 (NIH); 2U19AI089992-06A1 (NIH)
Record Dates: First submitted 2022-03-15; First posted 2022-03-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; Autoimmune Blistering Disease; B-Cell Deficiency
MeSH Terms: conditions — Multiple Sclerosis | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, peripheral blood mononuclear cells (PBMC), DNA, skin biopsies, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy control: Healthy controls Participants will receive COVID19 vaccination according to standard of care (any FDA approved vaccine). They will donate serial biospecimens before and after vaccination according to the study design.
  Interventions: Biological: COVID19 vaccine
- Disease control: Disease controls (individuals with a qualifying autoimmune condition, but not treated with any immunomodulator).
  Participants will receive COVID19 vaccination according to standard of care (any FDA approved vaccine). They will donate serial biospecimens before and after vaccination according to the study design.
  Interventions: Biological: COVID19 vaccine
- B-cell depleted: Individuals with autoimmune disease (multiple sclerosis or autoimmune blistering disease) who are treated with B-cell depleting anti-CD20 monoclonal antibodies.
  Participants will receive COVID19 vaccination according to standard of care (any FDA approved vaccine). They will donate serial biospecimens before and after vaccination according to the study design.
  Interventions: Biological: COVID19 vaccine
- Other immunomodulator: Individuals with autoimmune disease (multiple sclerosis or autoimmune blistering disease) who are treated with a non-CD20 monoclonal antibody immunomodulator to treat their disease.
  Participants will receive COVID19 vaccination according to standard of care (any FDA approved vaccine). They will donate serial biospecimens before and after vaccination according to the study design.
  Interventions: Biological: COVID19 vaccine

INTERVENTIONS:
Biological: COVID19 vaccine — All participants receive one or more FDA-authorized COVID19 vaccinations according to standard of care and current medical recommendations. The intervention is not specifically administered as part of the study.

SUMMARY:
The purpose of this study is to understand the immune response to coronavirus disease-19 (COVID-19) vaccination in patients on B-cell depleting therapies (BCDT) over time, which in the future may help to inform clinical decision making in this patient population.

DETAILED DESCRIPTION:
This will be a prospective, observational cohort study consisting of individuals with autoimmune diseases who are undergoing treatment with anti-CD20 medications at the time they receive a vaccine against COVID-19. Control groups will include healthy individuals, individuals with autoimmune diseases on other immunomodulators, and individuals with autoimmune diseases not on immunotherapy.

Participants will undergo serial blood draws and saliva collections at prespecified time points surrounding vaccination. A subset of agreeable participants will undergo skin biopsy within days of the first vaccination, with the option to repeat skin biopsy after the second vaccination. Additional blood, saliva and skin biopsy specimens may be obtained after booster vaccinations or after known COVID19 infections .

Specimens collected will be used for studies aimed at (1) understanding the pathobiology of neurologic/inflammatory/immune diseases and the immunologic response to COVID-19 vaccination, (2) identifying how and why treatments used for neurologic/immune diseases may impact the effectiveness of vaccination, and (3) identifying dermatologic manifestations of the immunologic response to the COVID-19 mRNA vaccine.

The investigators are investigating both the production of antibodies against the virus over time and deeply interrogating the T-cell response to vaccination using methods that measure T-cell reactivity to the COVID-19 virus, including single cell RNA sequencing.

ELIGIBILITY:
Subjects with neurologic/immunologic condition:

* at least 18 years of age
* Known diagnosis of autoimmune neurologic disease (e.g. multiple sclerosis (MS), neuromyelitis optica, myelin oligodendrocyte glycoprotein (MOG) -associated disorder) or autoimmune blistering disease (AIBD).
* EITHER:

  * Treated with an anti-CD20 (rituximab, ocrelizumab) medications for >6 months at the time of vaccination (B-cell depletion therapy, BCDT)
  * On no immunomodulatory therapy for their autoimmune condition for >6 months at the time of vaccination
  * Treated with a non-BCDT immunotherapy
* No relapse of neurologic/immunologic disease for >6 months prior to the time of enrollment
* Subject is eligible and willing to receive COVID-19 vaccination in accordance with local and national guidelines, or subject intends to receive booster COVID-19 vaccination in accordance with recommendations from their primary medical team.
* No active skin condition (e.g. open sores) preventing blood draw

Healthy Controls:

* at least 18 years of age
* No evidence of neurological/immunologic disease/illness/condition
* Subject is eligible and willing to receive COVID-19 vaccination in accordance with local and national guidelines, or subject intends to receive booster COVID-19 vaccination in accordance with recommendations from their primary medical team.
* No active skin condition (e.g. open sores) preventing blood draw/skin biopsy

Exclusion Criteria:

* Use of high dose steroids for treatment of neurologic/immunologic disease within 1 month of COVID-19 vaccination
* Anti-CD20 B-cell depleting therapy infused within 2 weeks of first study visit
* Inability to comply with the requirements of the protocol, in the opinion of the primary investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be four groups of participants overall:
  * Patients with autoimmune neurologic/autoimmune blistering disease (AIBD) who are on B-cell depleting therapy (anti-CD20 monoclonal antibodies)
  * Patients with autoimmune neurologic/AIBD who are on other types of immunomodulators
  * Patients with autoimmune neurologic/AIBD who are untreated
  * Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in coronavirus disease 19 (COVID19) antibody titers over time | Baseline, 2 weeks post vaccine 1, pre-vaccine 2, 1 week post vaccine 2, 6 months post vaccine 2; pre- and 2 week post any additional vaccines
  COVID 19 spike and neutralizing antibody titers will be monitored serially
Change in severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) specific T-cell activation over time | Baseline, 2 weeks post vaccine 1, pre-vaccine 2, 1 week post vaccine 2, 6 months post vaccine 2; pre- and 2 week post any additional vaccines
  Flow cytometry characterizing immunophenotype of SARS-CoV2 specific T cells

SECONDARY OUTCOMES:
Skin biopsy analysis | 7 days post vaccine 1; 7 days post vaccine 2; 4 days post booster (all timepoints optional)
  Histologic and immunologic characterization of skin biopsy specimens, comparing vaccinated to unvaccinated arm, at one or more timepoints post-vaccination
Measurement of COVID19 antibodies in saliva | Baseline, 2 weeks post vaccine 1, pre-vaccine 2, 1 week post vaccine 2, 6 months post vaccine 2; pre- and 2 week post any additional vaccines
  Descriptive assessment of whether COVID antibodies can be detected in saliva at any time point
Immune analysis | Baseline, 2 weeks post vaccine 1, pre-vaccine 2, 1 week post vaccine 2, 6 months post vaccine 2; pre- and 2 week post any additional vaccines
  Deep immunologic assessment (flow cytometry, single cell RNA sequencing) of blood specimens; descriptive analysis at each timepoint with comparisons over time will be performed.
Changes in patient reported outcomes: COVID history | Baseline, 2 weeks post vaccine 1, pre-vaccine 2, 1 week post vaccine 2, 6 months post vaccine 2; pre- and 2 week post any additional vaccines
  Subjective reports of vaccination-associated symptoms and COVID risk factors (COVID-19 survey)
Change in patient reported outcomes: patient reported disability steps | Baseline, 2 weeks post vaccine 1, pre-vaccine 2, 1 week post vaccine 2, 6 months post vaccine 2; pre- and 2 week post any additional vaccines
  Subjects will complete Patient Derived Disability Step score
Change in patient reported outcomes: overall symptoms | Baseline, 2 weeks post vaccine 1, pre-vaccine 2, 1 week post vaccine 2, 6 months post vaccine 2; pre- and 2 week post any additional vaccines
  SymptoMS screening questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Erin Longbrake, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
Sequencing data will be made publicly available upon publication of the study. Other study related data will be made available upon request and presentation of an appropriate research plan by qualified researchers

DOCUMENTS (1):
  • Informed Consent Form (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT05286242/ICF_000.pdf